CLINICAL TRIAL: NCT05988112
Title: Locoregional Recurrence After Radiotherapy in Breast Cancer Patients Based on Molecular Subtypes
Brief Title: Locoregional Recurrence of Breast Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amira Ali Fekry Mohamed, Assistant lecturer, Assiut University
Other Study IDs: Amira Ali
Record Dates: First submitted 2023-08-04; First posted 2023-08-14 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Locoregional Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
our study will be retrospective on breast cancer patients to detect relation between the locoregional recurrence of breast cancer after radiotherapy and the molecular subtypes

DETAILED DESCRIPTION:
Having replaced lung cancer as the most common cancer globally, breast cancer today represent 1 in 8 cancer cases and a total of 2.3 million new cases in both sexes .

It Represents a quarter of all cancer cases in females, and it was the most commonly diagnosed cancer in women in 2020 , its burden has been growing in many parts of the world, particularly in transitioning countries . An estimated 685,000 women died from breast cancer in 2020, corresponding to 16% or 1 in every 6 cancer deaths in women.

In Egypt, it constitutes 33% of female cancer cases and more than 22,000 new cases diagnosed each year .

Treatment Strategies include Surgery, Chemotherapy ,Radiotherapy, Endocrinal (Hormonal) Therapy & Biological Therapy , according to stages and molecular subtypes

A majority of breast cancer patients undergoing surgical excision will receive radiotherapy as a local treatment, which will reduce local and regional recurrence (LRR), further elevating survival.

Slightly over 50% of women with early-stage breast cancer remain disease free for at least 10 years, but recurrences continue to occur long after primary diagnosis.

Several multigene molecular assays are currently under investigation to accurately identify patients with unfavorable prognosis .However, considering the lack of cost-effectiveness of these detection approaches, they are not easily applied on a large scale, especially in less developed countries. In contrast, immunohistochemical (IHC) staining profile is a cost-effective and popular surrogate.Based on IHC staining profiles, St Gallen International Breast Cancer Conference in 2013 classified breast cancer into four subtypes: Luminal A, Luminal B, HER2-positive, and triple-negative breast cancer (TNBC). This classification system has been widely used in clinical decision-making for the systemic management of breast cancer.

This classification depend on presence or absence of estrogen receptor (ER), progesterone receptor (PR), human epidermal growth factor (Her2) and Ki 67 as luminal A is positive for ER &PR, negative for Her2 with low Ki67, luminal B is ER positive, PR & Her2 may be positive or negative but with high Ki67, Her2 is ER &PR negative with Her2 positive, Triple negative (TN) is ER & PR & Her2 negative with high Ki67, with no benefit of hormonal or anti Her2 therapy.

Few studies done showed that Luminal A and B subtypes are generally associated with lower risks of regional nodal involvement at diagnosis and tend to have a more indolent evolution as compared with the other subtypes. Several retrospective studies have shown lower rates of LRR in luminal A as compared with the other subtypes, among whom luminal B is considered as intermediate risk with rates ranging between 1.5 and 8.7% and peak incidence during the first 5 years .

For HER2-positive patients, there are two distinct periods. In studies in which patients were not treated with HER2-targeted therapy, LRR rates ranged between 4 and 15% .

More recently, trastuzumab have positively modified the natural course of this BC subtype. patients with HER2-positive tumors who underwent surgery and received trastuzumab had LRR rate of 1.7%. This finding was supported by many studies, who also showed that trastuzumab treatment resulted in a decrease in LRR by 50%. This has also been observed in small tumors HER2-positive BC study after trastuzumab .

The TNG subtype was associated with increased LRR rates, after breast conservation and mastectomy (3-17%). Moreover, after the diagnosis of an LRR, the TNG subtype is associated with a high incidence of distant metastases .

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Male or female
* Histological proven breast cancer (IDC / ILC)
* with known receptor status
* Patient did mastectomy or breast conservative surgery +/- lymph node dissection .
* received radiotherapy
* on regular follow up

Exclusion Criteria:

* Metastatic from the start (stage 4)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients diagnosed with breast cancer in clinical oncology department , Assuit university hospital
Sampling Method: Non-Probability Sample
Enrollment: 265 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Determine Local & regional recurrence according to different molecular subtypes. | within 5 years from diagnosis
  radiologically or with re biopsy
- 5-year free survival | within 5 years from diagnosis
  radiologically

SECONDARY OUTCOMES:
Metastasis-Free Survival | within 5 years from diagnosis
  radiologically